CLINICAL TRIAL: NCT02902796
Title: Randomized Controlled Cross Over Study to Compare the Efficacy of 1000 Hertz (Hz), Burst, and Standard Spinal Cord Stimulation in Chronic Axial Pain Relief
Brief Title: Comparison of 1000 Hertz (Hz), Burst, and Standard Spinal Cord Stimulation in Chronic Pain Relief
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Center for Clinical Research, Winston-Salem, NC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: IIR-2016-01
Record Dates: First submitted 2016-08-31; First posted 2016-09-16 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2018-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group A (Active Comparator): Group A will consist of sequence of treatment with 3 stimulation modes. They are, in order, 1000 hertz, standard, and burst stimulation. Each stimulation modes will last 3 weeks, with 4 days of wash off between them. Each group treatments will take about 3 months, and subject will cross over into the other treatment group. Burst stimulation sends packets of electrical pulses, composed of pulse and packet frequency. 1000 hertz stimulation delivers tonic, sub perception stimulation. The standard stimulation mode, which will serve as the control, will be below 100 hertz, and its pulse strength will be above threshold, where patients will feel the tingling from the electrical pulses generated by the spinal cord stimulator.
  Interventions: Device: Spinal cord stimulator
- Treatment group B (Active Comparator): Group B will consist of sequence of treatment with 3 stimulation modes. They are, in order, burst stimulation, standard, and 1000 hertz. Each stimulation modes will last 3 weeks, with 4 days of wash off between them. Each group treatments will take about 3 months, and subject will cross over into the other treatment group. Burst stimulation sends packets of electrical pulses, composed of pulse and packet frequency. 1000 hertz stimulation delivers tonic, sub perception stimulation. The standard stimulation mode, which will serve as the control, will be below 100 hertz, and its pulse strength will be above threshold, where patients will feel the tingling from the electrical pulses generated by the spinal cord stimulator.
  Interventions: Device: Spinal cord stimulator

INTERVENTIONS:
Device: Spinal cord stimulator — Spinal cord stimulator will be programmed to deliver, according to the randomization status of the patient, burst, 1000 hertz, and standard stimulation during each treatment group.

SUMMARY:
A randomized controlled with cross over study compares efficacy of burst stimulation, 1000 hertz stimulation, and standard stimulation in an non-superiority trial. The study duration is approximately 24 weeks and each stimulation modes will last for approximately 3 weeks with approximately 4 days of wash off in between.

DETAILED DESCRIPTION:
Study will enroll 22 patients for the purpose of evaluation of efficacy of burst stimulation, 1000 hertz frequency stimulation or standard stimulation in patients who have a spinal cord stimulators implanted. Each patients will be randomized to either group A or B, where each groups consists of Burst, standard, and 1000 hertz frequency stimulation or vice versa with wash off period in between. The duration for each stimulation modes will be approximately 3 weeks, with approximately 4 days of wash off prior to starting the new stimulation mode and in between stimulation modes. Treatment duration for each groups will last about 3 months or less, and with cross over total duration of the study is about 6 months in total.

During the trial there will be 13 visits. The first visit will consist of screening visit activities and once the eligibility of the subjects are confirmed, they will be randomized and they can start the study immediately and begin their wash off period. After the initial visit/ randomization visit, there will be 12 follow up visits. At each visit, patients will be assessed for their pain, disability index, and their perception of their painful condition, as well as any adverse events and changes of medication usage or lack there of. At the end of the study, the data will be pooled to look at the pain level, disability index, and patients perceived changes in their painful condition for each treatment groups (Burst stimulation, 1000 hertz stimulation and standard stimulation) to determine if subject experienced equivocal pain relief from all three stimulation modes.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years and older, and younger than 75 years of age.
* Subject has had a Precision Spectra, or Plus spinal cord stimulator system implanted for chronic painful condition.
* Subject continues to receive adequate pain relief with greater than or equal to 50% pain relief based on pre-trial and pre-implant pain assessment.
* Device age should not be less than 2 months old.
* Subject is willing to comply with all requirements of the study.

Exclusion Criteria:

* Subjects who are getting <50% pain relief on current SCS based on pre-trial and pre-implant pain assessment.
* Currently diagnosed with cognitive impairment, or exhibits any characteristic, that would limit study candidate's ability to assess pain
* Unstable medical or psychiatric illness
* Urine drug screen shows controlled substance/s not prescribed by the prescribers.
* Lifetime history of psychosis, hypomania, or mania.
* Epilepsy, or dementia
* Substance abuse in the last 6 months
* Pregnant or breastfeeding
* Not on contraception for those of childbearing age. (Barrier methods, oral contraception, hormone injections, or surgical sterilization)
* Treatment with investigational drug within 30 days of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
NPRS | 3 weeks, and 4 days
  Pain rating on 10 point digital scale for average, best, worst, during last week, and current pain level to be collected at each follow up visits. Collected data for each stimulation modes will be compared against each other to assess efficacy of 1000 hertz, and burst stimulation against each other and against the standard stimulation to look for differences in pain rating among three stimulation modes. Data comparison will occur at the end of the study, which is expected to last about 6 months.

SECONDARY OUTCOMES:
Oswestry Disability Index | 3 weeks, and 4 days
  Set of questionnaires designed to assess the level of disability in chronic pain patients. Each patients will be assessed with this questionnaires at each follow up visits. Collected data for each stimulation modes will be compared against each other to assess effects of 1000 hertz, and burst stimulation against each other and against the standard stimulation on Oswestry Disability Index, and changes if any.
Patients Global Impression of Change | 3 weeks, and 4 days
  Patient's assessment of the improvement or worsening of their painful condition during the study, and these will be collected at each follow up visits. Collected data for each stimulation modes will be compared against each other to assess effects of 1000 hertz, and burst stimulation against each other and against the standard stimulation on PGIC scores, and changes if any.
Preferability Survey | 3, and 6 months; at the completion of each treatment groups.
  subject preference of one stimulation program out of 3 received

CONTACTS AND LOCATIONS:
Overall Officials: James North, MD, Principal Investigator — The Center for Clinical Research
Locations (1):
- Jason Hong, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared. Only the pooled data will be shared with public and at the scientific meetings.

REFERENCES:
- [Background] Simpson BA. Spinal cord stimulation. Br J Neurosurg. 1997 Feb;11(1):5-11. doi: 10.1080/02688699746627. No abstract available. PMID 9156011
- [Background] De Ridder D, Vanneste S, Plazier M, van der Loo E, Menovsky T. Burst spinal cord stimulation: toward paresthesia-free pain suppression. Neurosurgery. 2010 May;66(5):986-90. doi: 10.1227/01.NEU.0000368153.44883.B3. PMID 20404705
- [Background] De Ridder D, Plazier M, Kamerling N, Menovsky T, Vanneste S. Burst spinal cord stimulation for limb and back pain. World Neurosurg. 2013 Nov;80(5):642-649.e1. doi: 10.1016/j.wneu.2013.01.040. Epub 2013 Jan 12. PMID 23321375
- [Background] Schu S, Slotty PJ, Bara G, von Knop M, Edgar D, Vesper J. A prospective, randomised, double-blind, placebo-controlled study to examine the effectiveness of burst spinal cord stimulation patterns for the treatment of failed back surgery syndrome. Neuromodulation. 2014 Jul;17(5):443-50. doi: 10.1111/ner.12197. Epub 2014 Jun 19. PMID 24945621
- [Background] De Ridder D, Vancamp T, Lenders MW, De Vos CC, Vanneste S. Is preoperative pain duration important in spinal cord stimulation? A comparison between tonic and burst stimulation. Neuromodulation. 2015 Jan;18(1):13-7; discussion 17. doi: 10.1111/ner.12253. Epub 2014 Oct 21. PMID 25334057
- [Background] Kriek N, Groeneweg G, Huygen FJ. Burst Spinal Cord Stimulation in a Patient with Complex Regional Pain Syndrome: A 2-year Follow-Up. Pain Pract. 2015 Jul;15(6):E59-64. doi: 10.1111/papr.12295. Epub 2015 Apr 10. PMID 25858033
- [Background] Crosby ND, Goodman Keiser MD, Smith JR, Zeeman ME, Winkelstein BA. Stimulation parameters define the effectiveness of burst spinal cord stimulation in a rat model of neuropathic pain. Neuromodulation. 2015 Jan;18(1):1-8; discussion 8. doi: 10.1111/ner.12221. Epub 2014 Aug 21. PMID 25145400
- [Background] Van Havenbergh T, Vancamp T, Van Looy P, Vanneste S, De Ridder D. Spinal cord stimulation for the treatment of chronic back pain patients: 500-Hz vs. 1000-Hz burst stimulation. Neuromodulation. 2015 Jan;18(1):9-12; discussion 12. doi: 10.1111/ner.12252. Epub 2014 Oct 22. PMID 25339436
- [Background] de Vos CC, Bom MJ, Vanneste S, Lenders MW, de Ridder D. Burst spinal cord stimulation evaluated in patients with failed back surgery syndrome and painful diabetic neuropathy. Neuromodulation. 2014 Feb;17(2):152-9. doi: 10.1111/ner.12116. Epub 2013 Sep 24. PMID 24655043
- [Background] De Ridder D, Lenders MW, De Vos CC, Dijkstra-Scholten C, Wolters R, Vancamp T, Van Looy P, Van Havenbergh T, Vanneste S. A 2-center comparative study on tonic versus burst spinal cord stimulation: amount of responders and amount of pain suppression. Clin J Pain. 2015 May;31(5):433-7. doi: 10.1097/AJP.0000000000000129. PMID 24977394
- [Background] Kriek N, Groeneweg JG, Stronks DL, Huygen FJ. Comparison of tonic spinal cord stimulation, high-frequency and burst stimulation in patients with complex regional pain syndrome: a double-blind, randomised placebo controlled trial. BMC Musculoskelet Disord. 2015 Aug 25;16:222. doi: 10.1186/s12891-015-0650-y. PMID 26303326
- [Background] Ito S, Sugiura T, Azami T, Sasano H, Sobue K. Spinal cord stimulation for a woman with complex regional pain syndrome who wished to get pregnant. J Anesth. 2013 Feb;27(1):124-7. doi: 10.1007/s00540-012-1462-y. Epub 2012 Aug 15. PMID 23011119
- [Background] Yoo HS, Nahm FS, Yim KH, Moon JY, Kim YS, Lee PB. Pregnancy in woman with spinal cord stimulator for complex regional pain syndrome: a case report and review of the literature. Korean J Pain. 2010 Dec;23(4):266-9. doi: 10.3344/kjp.2010.23.4.266. Epub 2010 Dec 1. PMID 21217892